CLINICAL TRIAL: NCT06000709
Title: Randomized, Double-blinded, Comparison Between Ultrasound-Guided Genicular Nerve Phenol Neurolysis and Intra-articular Steroid Injections
Brief Title: Comparison Between Ultrasound-Guided Genicular Nerve Phenol Neurolysis and Intra-articular Steroid Injections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Javier Webar, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS25899
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee; Chronic Knee Pain
Keywords: Phenol; Injections, Intra-Articular; Steroids; Nerve Block
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Methylprednisolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided Genicular Nerve Phenol Neurolysis (Experimental): One time injection of 1.5 mL of phenol 6% at 3 target locations: superomedial, superolateral and inferomedial genicular nerves
  Interventions: Drug: 6% aqueous phenol; Drug: Intraarticular Knee Placebo
- Ultrasound-guided Intraarticular Steroid Injection (Active Comparator): Intraarticular knee injection of 40 mg of methylprednisolone acetate in a volume of 5 mL of saline
  Interventions: Drug: MethylPREDNISolone 40 MG; Drug: Genicular Nerve Placebo

INTERVENTIONS:
Drug: 6% aqueous phenol — 1.5 mL of aqueous phenol will be injected at each target genicular nerve under ultrasound guidance
  Arms: Ultrasound-guided Genicular Nerve Phenol Neurolysis
Drug: MethylPREDNISolone 40 MG — 40 mg of methylprednisolone diluted in 5 mL of 0.9% normal saline will be injected inside the knee joint capsule under ultrasound guidance
  Arms: Ultrasound-guided Intraarticular Steroid Injection
Drug: Intraarticular Knee Placebo — Single injection 1.5 mL of 0.9% normal saline outside the knee joint capsule under ultrasound guidance
  Other Names: 0.9% normal saline
  Arms: Ultrasound-guided Genicular Nerve Phenol Neurolysis
Drug: Genicular Nerve Placebo — 1.5 mL of 0.9% normal saline will be injected subcutaneously at each target genicular nerve under ultrasound guidance
  Other Names: 0.9% normal saline
  Arms: Ultrasound-guided Intraarticular Steroid Injection

SUMMARY:
Genicular nerve neurolysis (GN) constitutes a relatively novel technique, whereby different chemical compounds (i.e. alcohol, phenol) are injected in close proximity to the genicular nerves of the knee joint, with the intention to exert a neurolytic effect by denaturing proteins resulting in Wallerian degeneration distal to the lesion. Based on the preliminary evidence and considering the potential benefits of the technique, we hypothesized that ultrasound-guided genicular chemical neurolysis with phenol is superior in terms of pain relief at 3 months, when compared to intra-articular steroid (IAS) injection.

DETAILED DESCRIPTION:
This study will allow us to determine if ultrasound-guided phenol genicular neurolys is superior to intra-articular steroid injection in terms of analgesia and functional outcomes, providing a more effective and long-lasting alternative for patients with chronic knee pain secondary to osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Severe knee pain for more than 6 months, defined as Numeric rating scale (NRS) score of 6 and greater, unresponsive to conservative medical treatment
* Radiological OA grade 2 to 4 (Kellgren-Lawrence scale)

Exclusion Criteria:

* Previous total knee replacement on the index knee
* Prior knee radiofrequency ablation on the index knee
* Connective tissue diseases with knee involvement (e.g. rheumatoid arthritis)
* Body mass index ≥ 40 kg/m2
* Uncontrolled coagulopathy, defined as supratherapeutic dose of anticoagulation medication
* Allergy to local anesthetics
* Unstable opioid consumption, defined as an increase >10% in dosage during the last 3 months prior to recruitment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores (Numeric Rating Scale) at 3 months | 3 months
  Knee pain intensity using Numeric Rating Scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Pain scores (Numeric Rating Scale) at baseline, 1 and 6 months | baseline, 1 month, 6 months
  Knee pain intensity using Numeric Rating Scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Proportion of patients experiencing a 50% or greater decrease in baseline knee pain scores (NRS) | 1 months, 3 months, 6 months
  Knee pain intensity using Numeric Rating Scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Brief Pain Inventory Score (BPI) | baseline, 1 month, 3 months, 6 months
  Functional activity measurement using the Brief Pain Inventory (short form)
WOMAC index | baseline, 1 month, 3 months, 6 months
  The WOMAC index consists of three subscales: pain, stiffness, and physical function (17 questions overall)
Incidence of adverse events | from injection up to 1 month after intervention
  Determined by the presence of hypoesthesia, paresthesia, puncture site hematoma, and worsening pain or infection

CONTACTS AND LOCATIONS:
Overall Officials: Javier Webar, MD, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walega DR, McCormick ZL. Chemical Neurolysis of the Genicular Nerves for Chronic Knee Pain: Reviving an Old Dog and an Old Trick. Pain Med. 2018 Sep 1;19(9):1882-1884. doi: 10.1093/pm/pny023. No abstract available. PMID 29514315
- [Background] Risso RC, Ferraro LHC, Nouer Frederico T, Peng PWH, Luzo MV, Debieux P, Sakata RK. Chemical Ablation of Genicular Nerve with Phenol for Pain Relief in Patients with Knee Osteoarthritis: A Prospective Study. Pain Pract. 2021 Apr;21(4):438-444. doi: 10.1111/papr.12972. Epub 2020 Dec 29. PMID 33277760
- [Background] Park Y, Lee SC, Nam HS, Lee J, Nam SH. Comparison of sonographically guided intra-articular injections at 3 different sites of the knee. J Ultrasound Med. 2011 Dec;30(12):1669-76. doi: 10.7863/jum.2011.30.12.1669. PMID 22124002
- [Background] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley D, Patel N, Choi D, Soloman M, Gupta A, Desai M, Buvanendran A, Kapural L. Prospective, Multicenter, Randomized, Crossover Clinical Trial Comparing the Safety and Effectiveness of Cooled Radiofrequency Ablation With Corticosteroid Injection in the Management of Knee Pain From Osteoarthritis. Reg Anesth Pain Med. 2018 Jan;43(1):84-91. doi: 10.1097/AAP.0000000000000690. PMID 29095245